CLINICAL TRIAL: NCT02430012
Title: Quality Measurement and Improvement Study of Surgical Coronary Revascularization: Secondary Prevention
Acronym: MISSION-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOST-2013BAI09B01-2
Record Dates: First submitted 2015-04-25; First posted 2015-04-29 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2015-06

CONDITIONS: Coronary Artery Bypass Grafting; Secondary Preventions
Keywords: coronary artery bypass grafting; quality improvement; secondary preventions

STUDY DESIGN:
Intervention Model Description: The study was a cluster randomized controlled trial to test the effectiveness of a smartphone-based multifaceted intervention. Sixty hospitals were randomized to the intervention group (n=30) or control group (n=30). Clinicians at intervention hospitals received multifaceted interventions (i.e., centralized training, evidenced-based checklists, and performance monitoring and feedback report) aimed at improving discharge prescription adherence, while those at control hospitals maintained routine practice.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor and data extractors were blind to the results of randomization
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): The intervention group will take the secondary prevention quality improvement strategies into implementation.
  Interventions: Behavioral: Quality improvement strategies
- Control group (No Intervention): The control goup will maintain the routine practice pattern.

INTERVENTIONS:
Behavioral: Quality improvement strategies — Training with guidelines of secondary preventions; determining improvement goals; tools (workflow posters and cards, checklists to inform the use of secondary prevention medications); periodical quality feedback report.
  Arms: Intervention group

SUMMARY:
The investigators have identified underuse of secondary prevention medications at discharge of patients underwent coronary artery bypass grafting (CABG) in China. The aim of this study is to develop series of quality improvement strategies focusing on secondary prevention medications for patients underwent CABG, and to evaluate their effectiveness and safety via a hospital-level cluster randomized clinical trial. The investigators established a network of 60 hospitals which have participated into Chinese Cardiovascular Surgery Registry and submitted 50 or more CABG surgeries already. The participating sites will be divided into intervention and control groups in a 1:1 ratio. The intervention group will undertake intervention of quality improvement strategies, while the control group will maintain the routine practice pattern. All hospitals will consecutively enroll and submit data of CABG during the enrollment period, estimated for 6 months. The prescribing rates of angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), beta-blockers, statins and aspirins will be compared between 2 groups.

DETAILED DESCRIPTION:
The investigators have identified underuse of secondary prevention medications at discharge of patients underwent coronary artery bypass grafting (CABG) in China. The aim of this study is to develop series of quality improvement strategies focusing on secondary prevention medications for patients underwent CABG, and to evaluate their effectiveness and safety via a hospital-level cluster randomized clinical trial. The investigators established a network of 60 hospitals which have participated into Chinese Cardiovascular Surgery Registry and submitted 50 or more CABG surgeries already. The participating sites will be divided into intervention and control groups in a 1:1 ratio. The intervention group will undertake intervention of quality improvement strategies, while the control group will maintain the routine practice pattern. All hospitals will consecutively enroll and submit data of CABG during the enrollment period of estimated 6 months. The prescription rates of ACEI, ARB, beta-blockers, statins and aspirins will be compared between 2 groups.

Before the enrollment period, the investigators have developed series of quality improvement strategies focusing on secondary prevention medications for patients underwent CABG, including training with guidelines of secondary preventions, determining improvement goals with participating sites, intervention tools (workflow posters and cards, checklists to inform the use of secondary prevention medications) and periodical quality feedback reports.

In the enrollment period, participating hospitals will be divided into intervention and control groups in a 1:1 ratio using minimization allocation.

The investigators will collect data on the prescription rates from central medical record abstraction, case report forms submitted by participating sites and checklists submitted by intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent CABG during the enrollment period in participating sites

Exclusion Criteria:

* Patients who die during hospitalization
* Patients who withdrawn from hospital against doctors' recommendations
* Patients who transfer out to other medical care institutions without discharge prescription

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10009 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09-18 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
statins use at discharge | 14 days on average (during hospitalization)
  Proportion of statins prescription at discharge among eligible patients

SECONDARY OUTCOMES:
ACEI/ARBs use at discharge | 14 days on average (during hospitalization)
  Proportion of β-blockers prescription at discharge among eligible patients
β-blockers use at discharge | 14 days on average (during hospitalization)
  Proportion of β-blockers prescription at discharge among eligible patients
aspirins use at discharge | 14 days on average (during hospitalization)
  Proportion of aspirins prescription at discharge among eligible patients

OTHER OUTCOMES:
education on smoking cessation at discharge | 14 days on average (during hospitalization)
  Proportion of education on smoking cessation at discharge among eligible patients
education on glycemic control at discharge | 14 days on average (during hospitalization)
  Proportion of education on glycemic control at discharge among eligible patients
education on moderate exercise at discharge | 14 days on average (during hospitalization)
  Proportion of education on moderate exercise at discharge among eligible patients
education on weight control at discharge | 14 days on average (during hospitalization)
  Proportion of education on weight control at discharge among eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, PhD, Study Director — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, People's Republic of China; Zhe Zheng, MD, PhD, Principal Investigator — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, People's Republic of China
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China